CLINICAL TRIAL: NCT04929782
Title: Clinical Evaluation of Giomer and Resin-based Fissure Sealants Performed in Permanent Molar Teeth Affected by Molar-Incisor Hypomineralization
Brief Title: Clinical Evaluation of Giomer and Resin-based Fissure Sealants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Beste Ozgur, Asst. Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUDHF-MIH-fissureselant
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Molar Incisor Hypomineralization
Keywords: molar incisor hypomineralization; giomer fissure sealants; resin sealants; adhesion
MeSH Terms: conditions — Molar Hypomineralization; Tissue Adhesions

STUDY DESIGN:
Intervention Model Description: Two intervention groups and split-mouth design
Who Masked: Outcomes Assessor
Masking Description: The follow-up evaluations by using the modified United States Public Health Service (USPHS) criteria were completed independently by two calibrated investigators who were blinded to the groups and a forced consensus was sought in any case of disagreement.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resin-based sealant (Active Comparator): A dental isolation device was used (Mr. Thisty One Step, Zirc Dental, Buffalo, MN, USA) and the treatments were conducted by one operator according to following steps; Group 1: Etching with 37% phosphoric acid for 30 s (i-GEL N, i-dental, Lithuania), rinsing for 30 s with air-water spray and drying with oil-free air for 15 s, resin sealant (Conceal F, SDI, Australia) application into the occlusal and buccal/palatal pits and fissures with direct placement syringe system and light curing with 460-500 nm wavelength halogen light unit (Hilux Dental Curing Light Unit 250, Benlioğlu Dental Inc, Turkey) for 20s on each surface.
  Interventions: Device: Resin-based sealant
- Giomer sealant (Active Comparator): Group 2: Self-etch primer (BeautiSealant Primer, Shofu, Japan) application to the occlusal and buccal/palatal pits and fissures with fine microbrush and waiting for 5 s, homogenizing the bond layer with gentle air stream for 5 s, giomer sealant application (BeautiSealant Paste, Shofu, Japan) with direct placement syringe system and light curing with 460-500 nm wavelength halogen light unit (Hilux Dental Curing Light Unit 250, Benlioğlu Dental Inc, Turkey) for 20 s on each surface.
  Interventions: Device: Giomer sealants

INTERVENTIONS:
Device: Resin-based sealant — Etching with 37% phosphoric acid for 30 s (i-GEL N, i-dental, Lithuania), rinsing for 30 s with air-water spray and drying with oil-free air for 15 s, resin sealant (Conceal F, SDI, Australia) application into the occlusal and buccal/palatal pits and fissures with direct placement syringe system and light curing with 460-500 nm wavelength halogen light unit (Hilux Dental Curing Light Unit 250, Benlioğlu Dental Inc, Turkey) for 20s on each surface.
  Other Names: Conceal F
  Arms: Resin-based sealant
Device: Giomer sealants — Self-etch primer (BeautiSealant Primer, Shofu, Japan) application to the occlusal and buccal/palatal pits and fissures with fine microbrush and waiting for 5 s, homogenizing the bond layer with gentle air stream for 5 s, giomer sealant application (BeautiSealant Paste, Shofu, Japan) with direct placement syringe system and light curing with 460-500 nm wavelength halogen light unit (Hilux Dental Curing Light Unit 250, Benlioğlu Dental Inc, Turkey) for 20 s on each surface.
  Other Names: BeautiSealant
  Arms: Giomer sealant

SUMMARY:
The objective of this research was to evaluate the clinical success of giomer and resin-based sealants applied in the first permanent molars (FPMs) affected by MIH.

DETAILED DESCRIPTION:
One-hundred FPMs with MIH which were indicated for non-invasive fissure sealant were selected in 39 children (between 6-12 years). Using a split mouth design, the FPMs were randomized into two groups; Group 1: resin sealant (Conceal F); Group 2: giomer sealant (BeautiSealant) and dental isolation device was used during the procedure (Mr. Thursty). Clinical evaluation was performed by two blinded examiners using the United States Public Health Service (USPHS) criteria to assess anatomical form, marginal adaptation, surface texture, marginal discoloration, retention and secondary caries at 1, 3, 6 and 12 months. Statistical analysis was performed using SPSS 20.0 software (IBM Corp., Chicago, IL, USA) and the level of significance was set at p<0.05. The association between independent variable (groups) and dependent variable (USPHS scores) was evaluated with Fisher's exact test. The crosstabulation of the categorical data regarding the groups were analyzed with chi-square test or Fisher's exact test. The Log-rank test and Kaplan-Meier analysis were used to calculate and compare the cumulative survival rates of the sealants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children, aged 6-12 years, who attended the pediatric dentistry clinic regular dental examination
* Cooperative children diagnosed with MIH according to European Academy of Paediatric Dentistry (EAPD) criteria
* Presenting at least two FPMs that were fully erupted and indicated for non-invasive fissure sealant.
* The FPMs with white, yellow or brown lesions, indicating mechanical and chemical alteration of the enamel and increased caries risk

Exclusion Criteria:

* Children having hypomineralized FPMs with post-eruptive breakdown, cavitated carious lesions, restorations or fixed orthodontic appliances
* Enamel defect due to a condition other than MIH

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Clinical performance evaluation using USPHS Criteria | 12 months
  Clinical evaluation was performed by two blinded examiners in accordance with the modified-USPHS criteria, to assess anatomic form, marginal adaptation, surface texture, marginal discoloration, retention and secondary caries at 1, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weerheijm KL, Jalevik B, Alaluusua S. Molar-incisor hypomineralisation. Caries Res. 2001 Sep-Oct;35(5):390-1. doi: 10.1159/000047479. No abstract available. PMID 11641576
- [Background] Fragelli CMB, Souza JF, Bussaneli DG, Jeremias F, Santos-Pinto LD, Cordeiro RCL. Survival of sealants in molars affected by molar-incisor hypomineralization: 18-month follow-up. Braz Oral Res. 2017 Apr 27;31:e30. doi: 10.1590/1807-3107BOR-2017.vol31.0030. PMID 28489117
- [Background] Lygidakis NA, Dimou G, Stamataki E. Retention of fissure sealants using two different methods of application in teeth with hypomineralised molars (MIH): a 4 year clinical study. Eur Arch Paediatr Dent. 2009 Dec;10(4):223-6. doi: 10.1007/BF03262686. PMID 19995506
- [Derived] Elmokanen MA, Gad HMA. Retention rate of giomer S-PRG filler containing pit and fissure sealant applied with or without etching: a randomized clinical trial. BMC Oral Health. 2024 Nov 7;24(1):1356. doi: 10.1186/s12903-024-05096-7. PMID 39511504
- [Derived] Ozgur B, Kargin ST, Olmez MS. Clinical evaluation of giomer- and resin-based fissure sealants on permanent molars affected by molar-incisor hypomineralization: a randomized clinical trial. BMC Oral Health. 2022 Jul 5;22(1):275. doi: 10.1186/s12903-022-02298-9. PMID 35790955